CLINICAL TRIAL: NCT03993886
Title: A Study AnalyZing a NovEl Wearable SeNsor for Remote PatIent Health Monitoring
Acronym: ZENITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReThink Medical (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P 005; 5R44HL125001-03 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-06-21 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Chronic Kidney Diseases
Keywords: Hemodialysis
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — Fitness Trackers

STUDY DESIGN:
Intervention Model Description: Multi-Arm study with different patient populations evaluating the CorBand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Arm 1 (Other): Adult (≥ 18 years of age) ambulatory patients diagnosed with heart failure and/or undergoing cardiac management.
  Interventions: Device: CorBand; Other: ECG; Other: respiratory rate sensor
- Arm 2 (Other): Adult (≥ 18 years of age) patients undergoing chronic hemodialysis.
  Interventions: Device: CorBand; Other: Activity Monitor; Other: Bioimpedance spectrometer
- Arm 3 (Other): Adult (≥ 18 years of age) patients (i) implanted with the CardioMEMS HF device and (ii) diagnosed with heart failure and/or undergoing cardiac management.
  Interventions: Device: CorBand
- Arm 4 (Other): Adult (≥ 18 years of age) patients diagnosed with heart failure and/or undergoing cardiac management.
  Interventions: Device: CorBand

INTERVENTIONS:
Device: CorBand — The CorBand device is a wrist-worn biosensor measuring heart rate, heart rate variability, respiration rate, skin temperature, bioimpedance, and activity.
Other: Activity Monitor — commercially available accelerometer to be worn on wrist
  Arms: Arm 2
Other: Bioimpedance spectrometer — Commercially available bioimpedance monitor.
  Arms: Arm 2
Other: ECG — Commercially available electrocardiogram machine
  Arms: Arm 1
Other: respiratory rate sensor — Commercially available respiratory rate sensor.
  Arms: Arm 1

SUMMARY:
Evaluate the performance of the CorBand product when used to monitor patients.

DETAILED DESCRIPTION:
The goal of the study is to demonstrate the validity and reliability of the CorBand across a suite of six clinical measures by comparing the measurements to similar outputs of FDA cleared devices:

* CorBand heart rate and heart rate variability will be compared to an electrocardiogram.
* CorBand bioimpedance will be compared to recorded extracted fluid and a bioimpedance measurement device.
* CorBand respiration rate will be compared to an respiratory rate sensor.
* CorBand skin temperature will be compared to a skin temperature monitoring device.
* CorBand activity will be compared to an activity monitor.
* CorBand outputs will be compared to the outputs of the CardioMEMS system.

Device safety, comfort, and ease-of-use will also be evaluated as part of this study. Adverse events and serious adverse events will be documented throughout the study duration.

ELIGIBILITY:
INCLUSION:

Arm 1:

1. Subject is ≥ 18 years of age (legal age to give informed consent).
2. Subject is NYHA class I, II, III, or IV or undergoing cardiac management at the time of enrollment.
3. Willing and capable of participating in all study visits and complying with medication/treatment requirements associated with this clinical study at an approved clinical study center.

Arm 2:

1. Subject is ≥ 18 years of age (legal age to give informed consent).
2. Subject receives chronic hemodialysis.
3. Subject undergoes at least two hemodialysis sessions per week.
4. Willing and capable of participating in all study visits and comply with medication/treatment requirements associated with this clinical study at an approved clinical study center.

Arm 3:

1. Subject is ≥ 18 years of age (legal age to give informed consent).
2. Subject is implanted with the CardioMEMS HF device.
3. Subject is NYHA class I, II, III, or IV or undergoing cardiac management at the time of enrollment.
4. Willing and capable of participating in all study visits and complying with medication/treatment requirements associated with this clinical study at an approved clinical study center.

Arm 4:

1. Subject is ≥ 18 years of age (legal age to give informed consent).
2. Subject is NYHA class I, II, III, or IV or undergoing cardiac management at the time of enrollment.
3. Subject is stabilized during (and not yet discharged from) a hospitalization for exacerbation of symptomatic heart failure or a clinic visit for symptomatic heart failure associated with unscheduled treatment with IV diuretics.
4. Willing and capable of participating in all study visits and complying with medication/treatment requirements associated with this clinical study at an approved clinical study center.

EXCLUSION:

1. The subject is unable or refuses to sign the informed consent.
2. Subject is pregnant or planning to become pregnant during the study.
3. A life expectancy of less than 6 months per clinician discretion.
4. Subject has an implanted pacemaker or pacing device (Arm 1 and Arm 2 only).
5. Poor healthcare literacy that would prevent the subjects from using the CorBand and/or completing questionnaires.
6. Physical or mental impairment preventing use of the CorBand or compliance with study requirements.
7. Material sensitivity to wearable devices, including the CorBand device.

   Additional Exclusion Criteria for Arm 4 Only:
8. Home use of intravenous continuous inotropes or planned outpatient weekly inotrope infusions.
9. Subject has been implanted with a ventricular assist device.
10. Subject is listed on heart transplant list.
11. Subject has a glomerular filtration rate (GFR) less than 30 mL/min.
12. Subject has uncontrolled hypertension defined as 160/100 mmHg on two consecutive readings taken 15 min apart after subject has been resting for 15 min.
13. Subject is undergoing or expected to undergo chronic hemodialysis (regularly scheduled sessions unrelated to a worsening heart failure event) during the study.
14. Subject is incompatible with CorBand (e.g., skin type resulting in poor data measurements).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Study Endpoint: Heart Rate | Through study completion, an average of 1 week
  To evaluate the accuracy of the heart rate data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)
Study Endpoint: Heart Rate Variability | Through study completion, an average of 1 week
  To evaluate the accuracy of the heart rate variability data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)
Study Endpoint: Respiration Rate | Through study completion, an average of 1 week
  To evaluate the accuracy of the respiration rate data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)
Study Endpoint: Activity | Through study completion, an average of 1 week
  To evaluate the accuracy of the activity (steps/movement) data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)
Study Endpoint: Skin Temperature | Through study completion, an average of 1 week
  To evaluate the accuracy of the skin temperature data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)
Study Endpoint: Bioimpedance (Extracellular fluid differences) | Through study completion, an average of 1 week
  To evaluate the accuracy of the bioimpedance (extracellular fluid differences) data collected by the CorBand compared to gold standard monitor. (No therapy or health outcomes will be evaluated. Data will assist in developing the decision model using the feature selection for the CorBand algorithm.)

OTHER OUTCOMES:
Incidence of investigational device related adverse events | Through study completion, an average of 1 week
  Adverse events and serious adverse events will be documented throughout the study duration.
Patient Experience | Through study completion, an average of 1 week
  Arm 2 and 3 Subjects will complete an end of study questionnaire to evaluate comfort and ease of use of the investigational device

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Kennedy, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Satellite Healthcare, San Jose, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Executive Summary: Heart Disease and Stroke Statistics--2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):447-54. doi: 10.1161/CIR.0000000000000366. No abstract available. PMID 26811276
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835